CLINICAL TRIAL: NCT05243251
Title: Olanzapine in Cancer Cachexia-Associated Anorexia: a Double-Blind Placebo-Controlled Randomized Clinical Trial
Brief Title: Olanzapine Anorexia Cachexia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Osama Ahmed, Demonstrator (Dr), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OlanCA
Record Dates: First submitted 2021-10-17; First posted 2022-02-17 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Anorexia
MeSH Terms: conditions — Anorexia | interventions — Olanzapine

STUDY DESIGN:
Intervention Model Description: This is a placebo-controlled double-blinded phase III randomized clinical trial. One hundred and sixty-four adult incurable cancer patients under treatment at Kasr Al-Ainy Center of Clinical Oncology and Nuclear Medicine (NEMROCK) - Kasr Al-Ainy School of Medicine - Cairo University during the period from December 2021 to September 2022.
  A written informed consent is to be obtained from all patients before entering the study. Then the investigators will give them dietary advice at baseline. Routine labs as complete blood count, liver, kidney function tests and CRP will be obtained to assess safety to start the drug and to assess its dose adjustment.
  Participants will be 1:1 randomized to the intervention (olanzapine) arm or the control (placebo) arm. Olanzapine will be given as oral 5 mg tablets (Zyprexa) and the placebo will be given in the form of tablets containing 300 mg of microcrystalline cellulose.
Who Masked: Participant, Investigator
Masking Description: We will prepare 82 jars containing the oral olanzapine tablets and similar 82 jars containing the placebo tablets. Each jar will have a unique number from 1 to 164. The jars will be prepared by Dr. Noha Abdel Razek, The Oncology Pharmacy Director at the department.
  The codes of the jars will be safeguarded till the end of the study at a closed cupboard at our clinic. The jars will be uncoded only at the end of the study by only one investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olanzapine (Active Comparator): 82 patients will receive olanzapine 5 mg daily at night for 4 weeks
  Interventions: Drug: Olanzapine 5 MG
- Placebo (Placebo Comparator): 82 patients will receive placebo for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olanzapine 5 MG — , Olanzapine (OLZ) is an atypical antipsychotic agent that blocks multiple neurotransmitters: dopamine at D1, D2, D3 and D4 brain receptors, serotonin at 5-HT2a , 5-HT2c, 5-HT3, and 5-HT6receptors, catecholamines at alpha 1 adrenergic receptors, acetylcholine at muscarinic receptors, and histamine at H1 receptors is suggested to have a valuable role in CAC
  Other Names: Zyprexa
  Arms: Olanzapine
Drug: Placebo — Tablets containing 300 mg of microcrystalline cellulose. It will be identical to the active drug
  Arms: Placebo

SUMMARY:
164 patients will be recruited..Adult patients diagnosed with incurable solid tumors and CCAA who presented to Kasr Al-Ainy Center of Clinical Oncology and Nuclear Medicine (NEMROCK) - Kasr Al-Ainy School of Medicine - Cairo University will be randomly distributed into 1:1..82 will receive Olanzapine 5 mg daily at night and 82 patients will receive placebo for 4 weeks. Primary outcome is Change in loss of appetite score from day 0 to day 7 of treatment and secondary outcomes change in body weight, change in loss of appetite score..and change in quality of life

DETAILED DESCRIPTION:
This is a placebo-controlled double-blinded phase III randomized clinical trial. One hundred and sixty-four adult incurable cancer patients under treatment at Kasr Al-Ainy Center of Clinical Oncology and Nuclear Medicine (NEMROCK) - Kasr Al-Ainy School of Medicine - Cairo University during the period from December 2021 to September 2022.

A written informed consent is to be obtained from all patients before entering the study. Then the investigators will give them dietary advice at baseline. Routine labs as complete blood count, liver,kidney function tests and CRP will be obtained to assess safety to start the drug and to assess its dose adjustment.

Participants will be 1:1 randomized to the intervention (olanzapine) arm or the control (placebo) arm. Olanzapine will be given as oral 5 mg tablets (Zyprexa) and the placebo will be given in the form of tablets containing 300 mg of microcrystalline cellulose.

• Method of randomization: The randomization sequence will be generated online by "Random.org".The investigators will use the sequence generator for numbers, where the minimum value is "1" and the maximum value is "164".

• Method of blinding:

The investigators will prepare 82 jars containing the oral olanzapine tablets and similar 82 jars containing the placebo tablets. Each jar will have a unique number from 1 to 164. The jars will be prepared by Dr.Noha Abdel Razek, the Oncology Pharmacy Direstor at the department.

The codes of the jars will be safeguarded till the end of the study at a closed cupboard at our clinic. The jars will be uncoded only at the end of the study by only one investigator.

• Assessment of compliance: Compliance will be assessed by pill count method at the end of the study period (day 28) and by patient reporting at days 7, 14 and 21 (Lam et al, 2015).

• Safety: A patient study card (or patient ID card) will be distributed to each participant. This card contains important information of the study drug, and includes the contact of the research staff coordinator. The patients will be instructed to carry this card with them all the time (just like they carry their identity card) and show it to the nurse/physician every time they visit a clinic or hospital. If they do not have the card or have lost it, they should ask for another one from the clinical trial coordinator.

The investigators will assess patients' mentality to exclude delirium using Mini Mental Scale (MMS) (Symptom Guidelines of Hospice Palliative Care Program, 2019).

Toxicity will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

9. Study outcomes:

* Primary outcome

  o Change in loss of appetite score from day 0 to day 7 of treatment with olanzapine 5 mg orally once daily at night: on the loss of appetite item of the ESAS-r.
* Secondary outcomes

  * Change in loss of appetite score from day 0 to days 14, 21 and 28: on the loss of appetite item of the ESAS-r.
  * Change in quality-of-life from day 0 to day 28: assessed using the Functional Assessment of Anorexia/Cachexia Therapy (FAACT) quality-of-life questionnaire.
  * Change in body weight from day 0 to day 28: using BF100 (Beurer Company).
  * Change in body mass index from day 0 to day 28.
  * Change in lean body mass from day 0 to day 28: by bioimpedence analysis using BF100 (Beurer Company).
  * Change in handgrip strength from day 0 to day 28: using JAMAR Digital Hand Dynamometer (Patterson Medical Company)(model 12-0604).
  * Change in fatigue from day 0 to day 28: using the fatigue item of the ESAS-r.
  * Change in CRP level from day 0 to day 28.
  * Adverse events: assessed weekly using the CTCAE version 5.

    10. Sample size: A sample size of 164 patients will be recruited to our study. Considering a 1.5-point change on the 0-10 loss-of-appetite scale of the ESAS to be of clinical importance (Del Fabbro et al, 2013) and a standard deviation of 2.9 (Blum et al, 2014), 63 evaluable patients are needed in each arm to detect a 1.5 points difference in the average change of anorexia score between the two arms with a two-sided 0.05 significance and 80% power. To compensate for 30% dropout rate and taking into consideration the non-parametric analysis of the primary endpoint, the plan is to recruit a total of 164 patients. Sample size calculation was done using G*Power Version 3.1.9.6. (Faul et al, 2009).

    11. 11- Statistical analysis plan Categorical variables will be expressed as number and percentage. A Chi-square test was used to determine the significance of difference in categorical variables between two or more groups.

The normality of continuous variables will be tested using Shapiro-Wilk test. Normally-distributed continuous variables will be expressed as mean and standard deviation, and abnormally-distributed as median and interquartile range. The significance of difference in normally distributed continuous variables between two groups will be tested using independent sample t-test; and for abnormally-distributed variables, Mann-Whitney U test will be used. Paired-samples t-test was used to test the difference in normally-distributed continuous variables at time intervals; and the Wilcoxon signed rank test for abnormally-distributed. All statistical tests will be two-sided and a p-value value <0.05 will be considered significant.

Per-protocol analysis of the 1ry outcome and other outcome measures at day 14 will include all patients who completed 14 days of treatment according to the protocol. Similarly, patients who completed 28 days of treatment according to the protocol will be included in per-protocol analysis at 28 days.

An intention-to-treat analysis of the 1ry outcome and other outcome measures at day 14 will be performed after imputation of missing values. Participants who withdrew from the study after randomization and before receiving a single dose of the intervention were excluded from the intention-to-treat analysis. Missing outcome values will be imputed using the k nearest neighbour (kNN) imputation method with a k value of 11. This will be done using the Visualization and Imputation of Missing Values (VIM) package (Templ et al, 201) of R software, version 4.0.5 (R Core Team 2021).

Statistical analysis was executed using MedCalc version 19.5.3 for Windows (MedCalc Software Ltd, Ostend, Belgium).

ELIGIBILITY:
Inclusion Criteria:

* o Age ≥ 18 years old at time of informed consent

  * Confirmed diagnosis of incurable solid tumor (cancer patients with incurable disease receiving anti-cancer therapy with palliative intent or best supportive care).
  * Loss of appetite score ≥ 4 on a 0 to 10 loss of appetite scale where 10 = worst possible lack of appetite as assessed by the Arabic version of Edmonton Symptom Assessment Scale (R/ESAS r) (ESAS-r, 2021).
  * Cachexia defined as "loss > 5% of body weight over the last 6 months" or "any degree of weight loss > 2 % associated with a body mass index (BMI) < 20" (Fearon et al, 2011).
  * Ability to take pills orally and not dependent on tube feeding (no oral mucosal inflammation, active dysphagia or gastrointestinal tract obstruction).
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
  * Ability to understand and communicate in Arabic and willingness to sign a written informed consent.
  * Patients were allowed to receive three-weekly regimens of anti-cancer treatment with palliative intent except those containing highly emetogenic chemotherapeutic (HEC) agents/regimens according to the American Society of Clinical Oncology (Hesketh et al, 2020).
  * Clinically-predicted survival of > 3 months.
  * Normal organ function (creatinine ≤2× upper limit of normal, bilirubin ≤2; upper limit of normal).

Exclusion Criteria:

* o Weight gain for known cause, e.g. oedema or ascites.

  * Treatment with other antipsychotic agents during the past 30 days.
  * Hypersensitivity to olanzapine.
  * Premenopausal women with childbearing potential with a positive serum B-HCG pregnancy test.
  * Inability to maintain oral intake.
  * Central nervous system disease (e.g., brain metastases, seizure disorder, schizophrenia, bipolar disorder, dementia or delirium).
  * Patients on supplements or medications with potential appetite-stimulating activity, such as megestrol acetate, corticosteroids, or thalidomide.
  * Patients unwilling or unable to comply with the protocol.
  * Nausea and/or vomiting score >3 on a 0 to 10 scale where 10 = extreme nausea/vomiting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2021-12-25 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
appetite score | 1 week
  Change in loss of appetite score from day 0 to day 7 of treatment with olanzapine 5 mg orally once daily at night: on the loss of appetite item of the ESAS-r. Where 0 is no loss of appetite and 10 worst appetite ever.

SECONDARY OUTCOMES:
appetite score | weekly till week 4
  o Change in loss of appetite score from day 0 to days 14, 21 and 28: on the loss of appetite item of the ESAS-r. Wher 0 is no loss of appetite and 10 worst appetite ever.
Change in quality-of-life | day 28
  o Change in quality-of-life from day 0 to day 28: assessed using the Functional Assessment of Anorexia/Cachexia Therapy (FAACT) quality-of-life questionnaire.
body weight | day 28
  Change in body weight from day 0 to day 28: using BF100 (Beurer Company).
body mass index | day 28
  Change in body mass index from day 0 to day 28.
handgrip strength | day 28
  o Change in handgrip strength from day 0 to day 28: using JAMAR Digital Hand Dynamometer (Patterson Medical Company)(model 12-0604).
lean body mass | day 28
  o Change in lean body mass from day 0 to day 28: by bioimpedence analysis using BF100 (Beurer Company).
Fatigue | day 28
  Change in fatigue from day 0 to day 28: using the fatigue item of the ESAS-r. Wher 0 is no fatigue and 10 is worst fatigue ever.
CRP | day 28
  Change in CRP level from day 0 to day 28.
Adverse events | weekly till day 28
  Adverse events: assessed weekly using the CTCAE version 5.

CONTACTS AND LOCATIONS:
Overall Officials: S Al Sirafy, Professor, Study Director — Kasr el einy school of medicine Cairo University
Locations (1):
- Kasr Al-Ainy Center of Clinical Oncology & Nuclear Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No